CLINICAL TRIAL: NCT04840901
Title: A Phase 1, Open-Label, Single-Dose Bioequivalence Study of Injections of Lebrikizumab Using a 2-mL Pre-Filled Syringe With Needle Safety Device and an Investigational 2-mL Autoinjector in Healthy Participants
Brief Title: A Study of Lebrikizumab (LY3650150) Administered by Two Different Devices in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17955; J2T-MC-KGBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lebrikizumab (Reference) - Pre-Filled Syringe with Needle Safety Device (Experimental): 2-milliliter (mL) (125 milligrams per milliliter [mg/mL]) Lebrikizumab administered subcutaneously (SC) via pre-filled syringe with needle safety device (PFS-NSD).
  Interventions: Drug: Lebrikizumab
- Lebrikizumab (Test) - Autoinjector (Experimental): 2-mL (125 mg/mL) Lebrikizumab administered SC via autoinjector (AI).
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC.
  Other Names: LY3650150

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, lebrikizumab, that gets into the blood stream and how long it takes the body to get rid of lebrikizumab (LY3650150) when given using either a pre-filled autoinjector (AI) or a pre-filled syringe with needle safety device (PFS-NSD). The safety and tolerability of lebrikizumab will also be evaluated. The study will last up to 102 days.

ELIGIBILITY:
Inclusion Criteria:

* Are Overtly healthy males or nonpregnant females of childbearing or non-childbearing potential as determined through medical evaluation.
* Agree not to donate blood or plasma until after the end of their participation in the study
* Have a body mass index (BMI) within the range 18.0 to 32.0 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Are females who are pregnant or lactating.
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have a history or presence of psychiatric disorders
* Show evidence of human immunodeficiency virus infection.
* Show evidence of hepatitis C and/or hepatitis B
* Medical history of allergic reaction to humanized monoclonal antibodies
* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Smoke more than 10 cigarettes per day or the equivalent including electronic cigarettes or are unable to abide by CRU smoking restrictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - QPS, Springfield, Missouri
  - Covance Dallas, Dallas, Texas
  - LabCorp CRU, Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD): 2-milliliters (mL) (125 milligrams per milliliter [mg/mL]) Lebrikizumab administered subcutaneously (SC) via pre-filled syringe with needle safety device (PFS-NSD).
- Lebrikizumab (Test) - Autoinjector (AI): 2-mL (125 mg/mL) Lebrikizumab administered SC via autoinjector (AI).
Period: Overall Study
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI)
Started | 123 | 119
Received at Least One Dose of Study Drug | 122 | 119
Completed | 118 | 117
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Moved | 1 | 0
Not completed — Unable to comply with study schedule | 0 | 1
Not completed — Screen Failure - Randomized but Did Not Receive Study Drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD): 2-mL (125 mg/mL) Lebrikizumab administered subcutaneously (SC) via pre-filled syringe with needle safety device (PFS-NSD).
- Total: Total of all reporting groups
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI) | Total
Number analyzed (Participants) | 122 | 119 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.6) | 44.1 (13.2) | 44.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 64 | 137
  Male | 49 | 55 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 30 | 50
  Not Hispanic or Latino | 102 | 88 | 190
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 27 | 55
  White | 91 | 90 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122 | 119 | 241

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lebrikizumab
Description: PK: Cmax of Lebrikizumab
Time Frame: Predose: Day 1, and Postdose: Days 3, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 99
Population: All participants who received a full dose of Lebrikizumab and had evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD): 2-mL (125 mg/mL) Lebrikizumab administered SC via pre-filled syringe with needle safety device (PFS-NSD).
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI)
Number analyzed (Participants) | 120 | 118
micrograms per milliliter (µg/mL) | 38.5 (31) | 41.9 (31)
Statistical Analysis 1: Comparison: Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) vs Lebrikizumab (Test) - Autoinjector (AI); Test type: Equivalence — PK parameters were powered to test equivalence with a power of 90% that the 90% confidence interval (CI) of the geometric mean ratio fall within 0.8 to 1.25 equivalence margin; ANCOVA; Ratio of Geometric LS Mean = 1.09, 90% CI 2-sided [1.03 to 1.16]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Lebrikizumab
Description: PK: AUC[0-∞] of Lebrikizumab
Time Frame: Predose: Day 1, and Postdose: Days 3, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 99
Population: All participants who received a full dose of Lebrikizumab and had evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day per milliliter (µg*d/mL)
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI)
Number analyzed (Participants) | 106 | 100
micrograms*day per milliliter (µg*d/mL) | 1340 (29) | 1450 (26)
Statistical Analysis 1: Comparison: Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) vs Lebrikizumab (Test) - Autoinjector (AI); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of Geometric LS Mean = 1.07, 90% CI 2-sided [1.02 to 1.14]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of Lebrikizumab
Description: PK: AUC[0-tlast] of Lebrikizumab
Time Frame: Predose: Day 1, and Postdose: Days 3, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 99
Population: All participants who received a full dose of Lebrikizumab and had evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*d/mL
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI)
Number analyzed (Participants) | 117 | 117
µg*d/mL | 1250 (28) | 1360 (25)
Statistical Analysis 1: Comparison: Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) vs Lebrikizumab (Test) - Autoinjector (AI); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of Geometric LS Mean = 1.09, 90% CI 2-sided [1.03 to 1.14]

ADVERSE EVENTS:
Time Frame: Up to 99 days
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) | Lebrikizumab (Test) - Autoinjector (AI)
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/119
Other Adverse Events (participants affected / at risk) | 39/122 | 26/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lebrikizumab (Reference) - Pre-Filled Syringe With Needle Safety Device (PFS-NSD) (N=122) | Lebrikizumab (Test) - Autoinjector (AI) (N=119)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 3 (3)
Injection site warmth (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Ulcer (General disorders) | 0 (0) | 1 (1)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginitis (Infections and infestations) | 0/73 (0) | 1/64 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 15 (18) | 7 (14)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/73 (0) | 1/64 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0/73 (0) | 2/64 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT04840901/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT04840901/SAP_001.pdf